CLINICAL TRIAL: NCT05561244
Title: Assessment of Weekly Monitoring Strategy of Capillary INR Versus Monthly Monitoring Strategy of Venous INR in Elderly Patients in a Nursing Home: Multicentre Randomised Cluster Trial.
Brief Title: Weekly Monitoring Strategy of Capillary INR Versus Monthly Monitoring Strategy of Venous INR in Elderly Patients in a Nursing Home.
Acronym: INR-CAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In the absence of patients meeting the selection criteria, the study was prematurely terminated. The average number of patients on VKAs per EHPAD has fallen sharply because of the development of direct oral anticoagulants and the Covid crisis.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-A00516-37
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation; Deep Vein Thrombosis; Stroke
Keywords: Atrial Fibrillation; Thrombosis; Stroke; Elderly
MeSH Terms: conditions — Atrial Fibrillation; Venous Thrombosis; Stroke; Thrombosis

STUDY DESIGN:
Intervention Model Description: This study is interventional, prospective, comparative, superiority, multicentric, randomised by cluster, in closed cohort.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CONTROL GROUP (No Intervention): Control group (n = 16 nursing homes, 64 patients): Patients will be monitored as usual using the Venous International Normalised Ratio strategy. Practices will not be changed (i.e. prospective observation of real-life practices; according to recommendations, at least 1 Venous International Normalised Ratio per month will usually be performed) and patients will not receive any supplementary intervention specific to the trial. A reminder of good International Normalised Ratio practices will be provided to nurses and prescribers.
- INTERVENTIONAL GROUP (Experimental): Intervention group (n = 16 nursing homes, 64 patients): Patients in the interventional group will be monitored using the capillary International Normalised Ratio strategy every week, and more often if the International Normalised Ratio is not in the therapeutic target. Venous International Normalised Ratio punctures will also be performed as described for the control group in order to calculate the Time in Therapeutic Range equivalently in both groups. Specific training in handling the device and the dose adjustment protocol will be provided to nurses and prescribers.
  Interventions: Device: Weekly monitoring using the capillary International Normalised Ratio strategy

INTERVENTIONS:
Device: Weekly monitoring using the capillary International Normalised Ratio strategy — Patients in the interventional group will be monitored using the capillary International Normalised Ratio strategy every week, and more often if the International Normalised Ratio is not in the therapeutic target. Venous International Normalised Ratio punctures will also be performed as described for the control group in order to calculate the Time in Therapeutic Range equivalently in both groups. Specific training in handling the device and the dose adjustment protocol will be provided to nurses and prescribers.
  Arms: INTERVENTIONAL GROUP

SUMMARY:
This primary care study aims to compare the "time in therapeutic range" (TTR) of two strategies for monitoring the international normalized ratio (INR) over 6 months in nursing homes. The population consists of frail elderly patients for whom Anti-Vitamin K treatments are frequent, and who are consequently more prone to embolic and hemorrhagic complications.

DETAILED DESCRIPTION:
Biological monitoring is essential to avoid strokes, deep vein thrombosis and hemorrhage. Generally speaking, this consists of a venous sampling for the international normalized ratio (INR), for which the therapeutic target is approximately 2.5 (tolerance range between 2 and 3) for atrial fibrillation (AF) and deep vein thrombosis (DVT). INR values below 2 indicate high risks of a stroke or DVT, whereas INR values over 3 refer to high risks of hemorrhage. INR monitoring requires monthly follow-ups or even more frequently if the HAS BLED score is ≥ 3.

One parameter used to evaluate the benefit/risk ratio is the "time in therapeutic range" (TTR), referring to the time spent within the INR therapeutic target (INR between 2 and 3 for patients with Atrial Fibrillation/ Deep Vein Thrombosis). It is calculated using the Rosendaal method. According to the "European Society of Cardiology" guidelines, the minimum threshold necessary for a good risk/benefit ratio is 70%. In other countries, it has been shown that the TTR is higher: 61% in Canada, 64.4% in Spain, 68.9% in Italy and 76.2% in Sweden. Moreover, TTR determines the benefit/risk ratio of the treatment, which means that patients with a TTR < 60% have more than 2% absolute total mortality per patient-year compared to patients with TTR > 60%.

As for the pilot study (Manuscript accepted in August 2019 in the Journal of Internal Medicine ), we expect approximately half the patients to be aged over 90. Patients will be recruited in nursing homes where they are monitored by nurses and care quality managers who are responsible for ensuring compliance with good clinical practices. This limits the risk of non-compliance with preanalytical venous INR conditions. Eighteen percent of subjects over 85 are treated with vitamin-K antagonists (VKA). For elderly patients with atrial fibrillation (AF) or deep venous thrombosis (DVT), stroke prophylaxis is a real clinical challenge. VKA treatments are indicated for the prevention of strokes in patients with Atrial Fibrillation, DVT or those who have received heart valve implants. VKAs have a narrow therapeutic range: if they are under-dosed, the risk of embolism (AVC and DVT) is high, whereas in the event of an overdose, the risk of bleeding is high. Given the annual incidence of severe hemorrhage (3-5%), the risk of a hemorrhage is their main side effect. The incidence of brain hemorrhages is 0.6 per 100 patient-years, for gastrointestinal bleeding it is 1.0 per 100 patient-years, and the risk of other serious bleeding is 1.4 per 100 patient-years. This risk of bleeding is usually assessed using the HAS-BLED score. The risk of hemorrhage is 4.2% per year in patients over 75 versus 1.7% per year for those under 75.

Following the results of a pilot study (manuscript accepted in the Journal of Internal Medecine), the hypothesis is that a weekly monitoring strategy for capillary INR should increase the TTR of nursing home patients by 12% compared to the usual monitoring by venous INR, resulting in a decrease of thrombotic or hemorrhagic events.

ELIGIBILITY:
Inclusion Criteria: The population corresponds to nursing homes patients treated with Vitamin K Antagonists for more than six months, because INRc cannot be used while anticoagulation treatment is being introduced.

* The patient or his/her trusted-person/legal representative/tutor signed the consent form
* The patient is an adult and lives in a nursing home
* The patient has been on treatment with Vitamin K Antagonists for more than six months
* The patient's target INR range is 2,5 [2-3] or 3 [2,5-3,5]
* The patient is affiliated to a health insurance program

Exclusion Criteria:

* The patient is participating in a Type 1 interventional study involving human beings (Jardé law).
* The patient is in an exclusion period determined by another study
* The patient is under safeguard of justice.
* It is not possible to give the patient (or his/her trusted-person/legal representative/tutor) informed information.
* The patient has a short life expectancy (< 1 month)
* The Karnofky index is ≤ 20%

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Interventional group : Time in Therapeutic Range using the capillary International Normalized Range weekly monitoring strategy | Day 0
  The CoaguChek INRange® device will be used. This small, portable monitoring medical device has already been used in several studies and can be used in hospital beds. After washing the patient's hands, the nurse will insert the strip test into the device, massaging the fingers and hand to activate blood circulation, and perform a capillary puncture using the lancet. An 8 μL drop of blood is required and must be deposited on the test strip less than 180 seconds after inserting the strip into the device and within 15 seconds after the start of blood drop formation. The International Normalized Ratio is displayed within one minute. When the nurse has the result, he/she will complete the VKA dose software (i.e. puncture number, strip number, current VKA type, current VKA dose, INRc value). The software will give the next puncture day and the correct VKA dose. If the INR > 4, there will be an alert and the nurse will have to contact the general practitioner for the rest of the procedure.
Interventional group : Time in Therapeutic Range using the capillary International Normalized Range weekly monitoring strategy | Month 6
  The CoaguChek INRange® device will be used. This small, portable monitoring medical device has already been used in several studies and can be used in hospital beds. After washing the patient's hands, the nurse will insert the strip test into the device, massaging the fingers and hand to activate blood circulation, and perform a capillary puncture using the lancet. An 8 μL drop of blood is required and must be deposited on the test strip less than 180 seconds after inserting the strip into the device and within 15 seconds after the start of blood drop formation. The International Normalized Ratio is displayed within one minute. When the nurse has the result, he/she will complete the VKA dose software (i.e. puncture number, strip number, current VKA type, current VKA dose, INRc value). The software will give the next puncture day and the correct VKA dose. If the INR > 4, there will be an alert and the nurse will have to contact the general practitioner for the rest of the procedure.
Control group : Time in Therapeutic Range using the venous International Normalized Range monthly monitoring strategy | Day 0
  The Time in Therapeutic Range will be measured as a percentage
Control group : Time in Therapeutic Range using the venous International Normalized Range monthly monitoring strategy | Month 6
  The Time in Therapeutic Range will be measured as a percentage

SECONDARY OUTCOMES:
Interventional group: venous thromboembolic events occurring during the 6-month monitoring period. | Day 0 to Month 6
  In the group being monitored weekly with the CoaguChek INRange® device, the number of venous thromboembolic events occurring during the 6-month monitoring period will be recorded.
Interventional group: haemorrhagic events occurring during the 6-month monitoring period. | Day 0 to Month 6
  In the group being monitored weekly with the CoaguChek INRange® device, the number of haemorrhagic events occurring during the 6-month monitoring period will be recorded.
Control group: venous thromboembolic events occurring with the monthly venous monitoring strategy. | Day 0 to Month 6
  The number of venous thromboembolic events occurring during the 6-month monitoring period will be recorded.
Control group: haemorrhagic events occurring with the monthly venous monitoring strategy. | Day 0 to Month 6
  The number of haemorrhagic events occurring during the 6-month monitoring period will be recorded.
Interventional group : Time in Therapeutic Range using the capillary International Normalized Range weekly monitoring strategy in patients ≤90. | Day 0
Interventional group : Time in Therapeutic Range using the capillary International Normalized Range weekly monitoring strategy in patients ≤90. | Month 6
Interventional group : Time in Therapeutic Range using the capillary International Normalized Range weekly monitoring strategy in patients >90. | Day 0
Interventional group : Time in Therapeutic Range using the capillary International Normalized Range weekly monitoring strategy in patients >90. | Month 6
Control group: Time in Therapeutic Range using the monthly venous monitoring strategy in patients ≤90. | Day 0
Control group: Time in Therapeutic Range using the monthly venous monitoring strategy in patients ≤90. | Month 6
Control group: Time in Therapeutic Range using the monthly venous monitoring strategy in patients >90. | Day 0
Control group: Time in Therapeutic Range using the monthly venous monitoring strategy in patients >90. | Month 6
Interventional group : Cost-consequences study on the weekly INRc monitoring strategy | Month 6
  Cost in terms of hospitalisations (due to haemorrhagic, ischemic and thromboembolic events) using the weekly INRc monitoring strategy will be studied including the cost of the device (equipment and consumables) from the public health insurance's perspective and the nursing time from the point of view of the health care institution.
Interventional group : Budget impact analysis on the weekly INRc monitoring strategy | Year 3
  Estimation of the financial consequences in terms of hospitalisations (due to haemorrhagic, ischemic and thromboembolic events) of adopting the new intervention in France
Control group : Cost-consequences study on the monthly venous monitoring strategy | Month 6
  Cost in terms of hospitalisations (due to haemorrhagic, ischemic and thromboembolic events) using the monthly venous monitoring strategy will be studied from the public health insurance's perspective and the nursing time from the point of view of the health care institution.
Control group : Budget impact analysis on the monthly venous monitoring strategy | Year 3
  An estimation will be made of the financial consequences in terms of hospitalisations (due to haemorrhagic, ischemic and thromboembolic events.

CONTACTS AND LOCATIONS:
Overall Officials: Chloé SIKIRDJI, Dr., Principal Investigator — CHU de Nîmes (NUH) Place du Pr. Debré 30029 NIMES Cedex9; Karen ZERBIB, Dr., Principal Investigator — EHPAD "Korian Mas de Lauze", 17, Chemin du puits de Louiset 30900 NIMES; Patrick DUTILLEUL, Dr., Principal Investigator — EHPAD Résidence "l'Accueil", 75 Rue Louis Aragon, 30600 VAUVERT; Alain BROUSSE, Dr., Principal Investigator — EHPAD "Les Jardins de l'Escalette",1 Avenue Marechal Foch 30700 UZES; Elodie MILLION, Dr., Principal Investigator — EHPAD Malbosc, 345 Avenue de Fes 34090 MONTPELLIER; Philippe SERAYET, Dr., Principal Investigator — EHPAD "Sophia la Capitelle", 57 Rue Henri Pitot 30840 MEYNES; Thierry CORNILLE, Dr., Principal Investigator — EHPAD "Docteur Henry Granet", 23 Chemin de la grave 30390 ARAMON +EHPAD "Les oliviers", 420 Chem. de Ceserac 30490 MONTFRIN; Gilles SEYLER, Dr., Principal Investigator — EHPAD "les Caprésianes",111 r. Alphonse Daudet 30210 CABRIERES, "Villa Rediciano", 6 r. du 19 Mars 1962, 30129 REDESSAN; Gil MEYRAND, Dr., Principal Investigator — EHPAD "Les Jasses", 155 Rue des Clapas 30730 FONS; Philippe VERNEDE, Dr., Principal Investigator — EHPAD "Jacques Saurin", Avenue des Loisirs 30190 MOUSSAC; Katia BRUNEL, Dr., Principal Investigator — EHPAD "Jean Lasserre", Chem. des Camisards 30360 EUZET; Georges ALVADO, Dr., Principal Investigator — EHPAD "Les Capitelles", Impasse de la Thebaide 30620 BERNIS; Christine DE TADDEO, Dr., Principal Investigator — EHPAD Serre-Cavalier - Sites 1 & 2, Rue Pitot Prolongée 30000 Nîmes; Marie-Hélène GRAS-JAEN, Dr., Principal Investigator — EHPAD ORPEA "Château notre dame", Pl. du Château 30730 PARIGNARGUES; Marc BORGHERO, Dr., Principal Investigator — EHPAD Samdo Rochebelle, 17 Rue des Châtaigniers 30100 ALES; Anne-Laure VITEAU, Dr., Principal Investigator — EHPAD "Les 5 sens Garons", Carieire dis Amourous 30128 GARONS; Abderrahmane ALOUI, Dr., Principal Investigator — EHPAD Korian "Les Meunières" Place Denfert Rochereau 34400 LUNEL; Pierre MERLE, Dr., Principal Investigator — EHPAD du Centre hospitalier de Langogne, Clos de la Tuilerie 48300 LANGOGNE; Marc DUPUIS, Dr., Principal Investigator — EHPAD Saint-Vincent de Paul,16 Rue de l'Égalité 30240 LE GRAU-DU-ROI; Julie LANO, Dr., Principal Investigator — EHPAD "Coté Canal", 116 Rue Jacques Cœur 30220 AIGUES-MORTES; Florence CHAPOUTOUT, Dr., Principal Investigator — EHPAD "La belle viste", 149 Rue du parc BP 2 34980 ST GELY DU FESC; Nicole GARCIA, Dr., Principal Investigator — EHPAD "Les monts d'Aurelle",Parc Euromedecine 1632 Rue St Priest 34097 MONTPELLIER CEDEX 5; Robert LE STUM, Dr., Principal Investigator — Maison de Retraite Protestante, 2252 Rte de Mende 34090 MONTPELLIER; Marie-Aude BONNEL, Dr., Principal Investigator — EHPAD "les Dominicaines",2 Rue du Thirondel 34190 GANGES; Adrien ROMARY, Dr., Principal Investigator — EHPAD "Résidence les Magnans", 85 Rue du Dix Neuf Mars 1962, 30520 SAINT-MARTIN-DE-VALGALGUES; Mélanie BADIN, Dr., Principal Investigator — 68 rue du charron 30310 VERGEZE; Murielle GLONDU-LASSIS, Dr., Principal Investigator — SCM Médicale St Bauzille de Putois 1193 avenue du chemin neuf 34190 ST BAUZILLE DE PUTOIS; Hermine SAGUY, Dr., Principal Investigator — 2 rue Ibn Sinaï Dit Avicenne 66330 Cabestany; Anne-Sophie ODOUL, Dr., Principal Investigator — 392 Boulevard Pedro de Luna 34070 MONTPELLIER; Victor LIVIOT, Dr., Principal Investigator — EHPAD Léon Bourgeois 1 Place du Puig Tarrous 66740 VILLELONGUE DELS MONTS; Philippe Roure, Dr., Principal Investigator — EHPAD La Pinède 110 chemin des cades 30310 Vergeze; Franck Raschilas, Dr., Principal Investigator — Centre Bellevue-CHU Montpellier 1 Pl. Jean Baumel 34090 Montpellier; Chloé Loeffler, Dr., Principal Investigator — EHPAD La Murelle Avenue de la Gare 34480 - LAURENS
Locations (33):
- France (33):
  - EHPAD " Coté Canal ", Aigues-Mortes, GARD
  - EHPAD "Samdo Rochebelle", Alès, GARD
  - EHPAD "Docteur Henry Granet", Aramon, GARD
  - EHPAD "Les Capitelles", Bernis, GARD
  - EHPAD Résidence "Les Caprésianes", Cabrières, GARD
  - EHPAD "Jean Lasserre", Euzet, GARD
  - EHPAD "Les Jasses", Fons, GARD
  - EHPAD "Les 5 sens Garons", Garons, GARD
  - EHPAD Saint-Vincent de Paul, Le Grau-du-Roi, GARD
  - EHPAD "Sophia la Capitelle", Meynes, GARD
  - EHPAD "Les oliviers", Montfrin, GARD
  - EHPAD "Jacques Saurin", Moussac, GARD
  - EHPAD "Ma Maison", Nîmes, GARD
  - EHPAD Serre-Cavalier Sites 1 and 2, Nîmes, GARD
  - Nîmes University Hospital, Place du Pr. Debré, Nîmes, Gard
  - EHPAD ORPEA "Château Notre Dame", Parignargues, GARD
  - EHPAD "Villa Rediciano", Redessan, GARD
  - EHPAD "Résidence les Magnans", Saint-Martin-de-Valgalgues, GARD
  - EHPAD "Les Jardins de l'Escalette", Uzès, GARD
  - EHPAD Résidence "l'Accueil", Vauvert, GARD
  - EHPAD Korian "Les Meunières", Lunel, HERAULT
  - EHPAD Malbosc, Montpellier, HERAULT
  - SCM Médicale St Bauzille de Putois, Saint-Bauzille-de-Putois, HERAULT
  - EHPAD "Les Dominicaines", Ganges, Hérault
  - Maison de Retraite Protestante, Montpellier, Hérault
  - EHPAD "Les Monts d'Aurelle", Montpellier, Hérault
  - EHPAD "La BELLE Viste", Saint-Gély-du-Fesc, Hérault
  - EHPAD du centre hospitalier de Langogne, Langogne, LOZERE
  - EHPAD La Murelle, Laurens
  - Centre Bellevue-CHU Montpellier, Montpellier
  - EHPAD "Korian Mas de Lauze", Nîmes
  - EHPAD La Pinède, Vergèze
  - EHPAD Léon Bourgeois, Vilallonga dels Monts

IPD SHARING:
Plan to Share IPD: No